CLINICAL TRIAL: NCT02484040
Title: Two-Week COurse Versus Conventionally Fractionated Preoperative Chemoradiotherapy In Locally Advanced Rectal Cancer (TwoArc Trial): A Phase III Randomized Clinical Trial
Brief Title: Two-week Course Versus Conventionally Fractionated Chemoradiotherapy in Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jong Hoon Lee (Other)
Responsible Party: Sponsor-Investigator, Jong Hoon Lee, Mr., Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TwoArc trial
Record Dates: First submitted 2015-06-17; First posted 2015-06-29 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Response to Toxin; Toxicity; Recurrence
Keywords: tumor response; toxicity; recurrence; chemoradiotherpy; rectum
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Two-week course arm (Experimental): Experimental arm receive 33 Gy in 10 fractions of radiation for 2 weeks with oral capecitabine.
  Two-week course of radiation, 33 Gy/10 fx and oral capecitabine, 825 mg/m2, bid
  Interventions: Radiation: Two-week course of radiation; Drug: Two-week course of radiation
- Conventional arm (No Intervention): conventionally fractionated radiation of 50.4 Gy/28 fx and 5-FU, 500 mg/m2 and leucovorin, 20 mg/m2 for 5 days, monthly or Capecitabine, 825 mg/m2, bid

INTERVENTIONS:
Radiation: Two-week course of radiation — 33 Gy in 10 fractions for 2 weeks
  Other Names: experimental arm
  Arms: Two-week course arm
Drug: Two-week course of radiation — oral capecitabine, 825mg/m2, bid
  Other Names: experimental arm
  Arms: Two-week course arm

SUMMARY:
The investigators compare two-week course of chemoradiation (33 Gy in 10 fractions with oral capecitabine) and conventional chemoradiation (50.4 Gy in 28 fractions with 5-FU and leucovorin) in this randomized trial.

DETAILED DESCRIPTION:
1.1 experimental arm Two-week course concurrent chemoradiotherapy

* Radiotherapy, 33 Gy/10 fractions for 2 weeks

  ↓↓↓↓↓ ↓↓↓↓↓ Radical surgery 6 weeks after completion of chemoradiotherapy D1----------------------D12
* Capecitabine 825 mg/m2, twice daily

1.2 control arm

Standard concurrent chemoradiotherapy (CRT)

* Radiotherapy, 50.4 Gy/28 fractions for 6 weeks

  ↓↓↓↓↓ ↓↓↓↓↓ ↓↓↓↓↓ ↓↓↓↓↓ ↓↓↓↓↓ ↓↓↓ Radical surgery D1--------------------------------------------------------------------------D38
* Bolus 5-FU, 400 mg/ m2 and leucovorin, 20 mg/ m2 during week 1 and 5
* Capecitabine, 825 mg/ m2, bid

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed adenocarcinoma;
2. distal margin of the tumor located < 10 cm from the anal verge;
3. cT3-4N0-2 classification as determined by magnetic resonance imaging (MRI) and/or endorectal ultrasonography (EUS);
4. no evidence of distant metastasis;
5. Karnofsky performance score over 70;
6. adequate bone marrow, liver, and renal function (leucocytes >4000/mm3, hemoglobin >10 g/dL, platelets >100,000/mm3; serum bilirubin <1.5 mg/dL, serum transaminase <2.5 times the upper normal limit; serum creatinine <1.5 mg/dL).

Exclusion Criteria:

1. Metastatic disease
2. No complete resection of tumor (R2)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Tumor response from stage II-III to stage 0-I | from clinical staging time to radical surgery date (about 3 months)
  Downstaging rate was evaluated by comparing pre-clinical and post-CRT pathological stages, and downstaging was defined as ypStage 0-I (ypT0-2N0M0)

SECONDARY OUTCOMES:
Toxicity (acute and chronic) | from radiation start to 3 years after radical surgery
  During the course of radiotherapy, patients were evaluated weekly to assess acute toxicity. Patients were also followed 2 and 4 weeks after completion of radiotherapy and until 3 years after curative surgery to assess toxicity. Toxicity are assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0).
Recurrence and survival | 3-year recurrence-free survival and 3-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hoon Lee, MD, Principal Investigator — St. Vincent's Hospital, The Catholic University of Kora
Locations (1):
- Lee Jong Hoon, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Lee JH, Kim JG, Oh ST, Lee MA, Chun HG, Kim DY, Kim TH, Kim SY, Baek JY, Park JW, Oh JH, Park HC, Choi DH, Park YS, Kim HC, Chie EK, Jang HS. Two-week course of preoperative chemoradiotherapy followed by delayed surgery for rectal cancer: a phase II multi-institutional clinical trial (KROG 11-02). Radiother Oncol. 2014 Jan;110(1):150-4. doi: 10.1016/j.radonc.2013.11.013. Epub 2014 Jan 7. PMID 24411228